CLINICAL TRIAL: NCT05306236
Title: Efficacy of Adding Low Level Laser Therapy to Postural Correction Exercises on Postnatal Sacroiliac Joint Pain
Brief Title: Efficacy of Adding LLL Therapy to Postural Correction Exercises on Postnatal SIJ Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, manal ahmed el-shafei mohamed, lecturer of physical therapy for women's health, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003492
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Sacroiliac Joint Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LLL therapy and postural correction ex (study group) (Experimental): study group will be treated by low level laser therapy and postural correction exercises
  Interventions: Other: LLL therapy , postural correction ex
- postural correction ex (control group) (Experimental): control group will be treated by postural correction exercises only
  Interventions: Other: LLL therapy , postural correction ex

INTERVENTIONS:
Other: LLL therapy , postural correction ex — study group: will receive low level laser therapy 2 sessions per week for 6 weeks in addition to posture correction exercises.
  control group: will be treated by posture correction ex only.

SUMMARY:
the purpose of the study will be to to examine the effect of low level laser therapy on pain and function disability in postnatal women with sacroiliac joint pain.

DETAILED DESCRIPTION:
Women are more susceptible to sacroiliac joint pain than men because the physiological changes associated with childbearing (e.g. pregnancy associated with weight gain, exaggerated lumber lordosis, hormone-induced ligamentous laxity and the mechanical trauma associated with childbirth) may result in sacroiliac joint pathology .

Low level laser is effective for treatment of various musculoskeletal pain disorders. It releases local neurotransmitters such as serotonin and endorphins. Additionally, the analgesic effect of LLLT is thought to be related to its anti-inflammatory action. Laser irradiations also relieve pain by alleviating and removing swelling and by increasing oxygenation of the tissues, thus results in reduction of the pain .

ELIGIBILITY:
Inclusion Criteria:

* Post natal women suffering from sacroiliac joint pain for at least 3 months.
* They should have moderate to severe pain in the sacroiliac joint region (visual analogue scale ≥ 4).
* They should have positive findings in at least three of five provocation sacroiliac joint tests (i.e., Patrick's sign, Gaenslen test, compression test, thigh thrust test and distraction test).
* Their age will range from 25 to 40 years old.
* Their Body mass index (BMI) will be ranged from 25 to 30 Kg /m2.
* They should not have any musculoskeletal disorders.

Exclusion Criteria:

* Lumber or hip joint pathology.
* Acute pelvic bacterial or viral infections or tumour.
* Taking nonsteroidal anti-inflammatory drugs, or hormonal treatments.
* Having positive straight leg raising test.

Ages: 25 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-04-30 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-07-28 (Actual)

PRIMARY OUTCOMES:
pain intensity | up to 2 months
  The pain intensity will be assessed through visual analogue scale (VAS) for both groups before and after the end of treatment program. Each woman will be asked to mark a point on the line between the extremes that related to her pain intensity.
pain pressure threshold | up to 2 months
  pressure algometer will be used to assess pain pressure threshold for both groups before and at the end of the study

SECONDARY OUTCOMES:
functional disability | up to 2 months
  oswestery disability index will be used to assess level of functional disability for both groups before and at the end of the study

CONTACTS AND LOCATIONS:
Locations (1):
- Manal Ahmed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF